CLINICAL TRIAL: NCT01076179
Title: KALETRA in Combination With New Substances (PROTEKT)
Brief Title: Kaletra in Combination With Antiretroviral Agents
Acronym: PROTEKT
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P11-021
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: Infection; Rilpivirine; CCR5 antagonists; Etravirine; Human Immunodeficiency Virus; Maraviroc; Safety and efficacy; Non nucleoside reverse transcriptase inhibitors (NNRTIs); Integrase inhibitors; Raltegravir; Kaletra
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Human Immunodeficiency Virus (HIV)-Infected Participants: HIV-infected participants on Kaletra and INIs or NNRTIs or CCR5 antagonists

SUMMARY:
The purpose of this study is to investigate the tolerability of Kaletra (lopinavir/ritonavir) in combination with new substances such as integrase inhibitors (INIs), C-C chemokine receptor type 5 (CCR5) antagonists, and new non-nucleoside reverse transcriptase inhibitors (NNRTIs), as there are many reasons (intolerability, complex resistant patterns or even personal reasons) which may result in a change from the daily clinical routine and lead to the use of a newly approved antiretroviral agent in combination with Kaletra.

DETAILED DESCRIPTION:
This study was designed as a non-interventional observational study. Kaletra was prescribed in the usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18years of age
* Written informed consent (authorization to the investigator to use and/or disclose personal and/or health data before entry into the KALETRA® post marketing observational study)
* HIV-1 infection
* Patients treated with KALETRA®, independent from their participation in this study
* Patients treated with novel antiretroviral therapy (for at least 8 weeks according to the study amendment), independent from their participation in this study

Exclusion Criteria:

* Hypersensitivity against Kaletra or other ingredients or INIs or NNRTIs or CCR5 antagonists
* Severe liver insufficiency
* No concommitant astemizole, terfenadine, oral midazolam, triazolam, cisapride, pimozide, amiodarone, ergotamine, dihydroergotamine, ergometrine, methylergometrine, vardenafil and/or St. John's wort

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample: HIV-positive patients
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2008-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Wittig, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-infected Participants: Human immunodeficiency virus (HIV)-infected participants on Kaletra and integrase inhibitors (INIs) or non nucleoside reverse transcriptase inhibitors NNRTIs) or C-C chemokine receptor type 5 (CCR5) antagonists
Period: Overall Study
Arm/Group | HIV-infected Participants
Started | 502
Completed | 501
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- HIV-infected Participants: HIV-infected participants on Kaletra and INIs or NNRTIs or CCR5 antagonists
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 431

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Adverse Events (Weeks 0-144), Per Event
Description: Percentage of overall number of adverse events experienced during Weeks 0-144 by adverse event type. Doctors asked participants for adverse events, grouped them into categories given in the electronic case report form (eCRF). The list of adverse events included in the eCRF were hypertriglyceridemia, hypercholesterolemia, low high density lipoprotein (HDL) cholesterol, high low density lipoprotein (LDL) cholesterol, hyperglycemia, hyperbilirubinemia, elevated aspartate aminotransferase (AST), elevated alanine aminotransferase (ALT), elevated gamma glutamyl transferase (γGT), elevated alkaline phosphatase, stomatitis, nausea, vomiting, diarrhea, abdominal pain, mood disorder, neurocerebellar disorder, headache, fatigue, fever, other (listed as 'not specified').
Time Frame: Weeks 0 to 144
Measure: Number; unit: percentage of adverse events
Units Other Than Participants: Adverse Events
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 501
Number analyzed (Adverse Events) | 3450
percentage of adverse events
  Hypertriglyceridemia | 13.8
  Hypercholesterolemia | 19.3
  Low HDL Cholesterol | 1.0
  High LDL Cholesterol | 4.4
  Hyperglycemia | 1.6
  Hyperbilirubinemia | 1.8
  Elevated AST | 3.4
  Elevated ALT | 4.6
  Elevated γGT | 6.3
  Elevated Alkaline Phosphatase | 1.5
  Stomatitis | 0.6
  Nausea | 3.1
  Vomiting | 1.2
  Diarrhea | 14.9
  Abdominal Pain | 3.1
  Mood Disorder | 5.2
  Neurocerebellar Disorder | 0.8
  Headache | 1.3
  Fatigue | 1.7
  Fever | 1.2
  Not Specified | 9.1

2. Primary Outcome: Prevalence of Adverse Events (Weeks 0-144), Per Participant
Description: Percentage of participants who experienced at least 1 adverse event during Weeks 0-144 by adverse event type. Doctors asked participants for adverse events, grouped them into categories given in the eCRF. The list of adverse events included in the eCRF were hypertriglyceridemia, hypercholesterolemia, low HDL cholesterol, high LDL cholesterol, hyperglycemia, hyperbilirubinemia, elevated AST, elevated ALT, elevated γGT, elevated alkaline phosphatase, stomatitis, nausea, vomiting, diarrhea, abdominal pain, mood disorder, neurocerebellar disorder, headache, fatigue, fever, other (listed as 'not specified').
Time Frame: Weeks 0 to 144
Measure: Number; unit: percentage of participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 501
percentage of participants
  Hypertriglyceridemia | 14.8
  Hypercholesterolemia | 17.8
  Low HDL Cholesterol | 3.0
  High LDL Cholesterol | 7.2
  Hyperglycemia | 2.8
  Hyperbilirubinemia | 2.8
  Elevated AST | 5.0
  Elevated ALT | 6.4
  Elevated γGT | 7.8
  Elevated Alkaline Phosphatase | 3.2
  Stomatitis | 2.0
  Nausea | 8.6
  Vomiting | 4.0
  Diarrhea | 27.3
  Abdominal Pain | 7.8
  Mood Disorder | 9.8
  Neurocerebellar Disorder | 2.2
  Headache | 4.0
  Fatigue | 4.6
  Fever | 4.0
  Not Specified | 28.5

3. Secondary Outcome: Change From Baseline in Absolute Cluster of Differentiation 4 (CD4) Cell Count
Description: Changes in participants' CD4 cell counts were assessed by measuring the change from Baseline in the number of CD4 cells at scheduled visits planned as part of routine care.
Time Frame: Baseline (Week 0) to Week 144
Population: Participants with an assessment at Baseline. Number analyzed=participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 500
cells/μL
  Change at Week 4: number analyzed (Participants) | 369
  Change at Week 4 | 54.0 (161.7)
  Change at Week 12: number analyzed (Participants) | 400
  Change at Week 12 | 64.6 (148.5)
  Change at Week 24: number analyzed (Participants) | 414
  Change at Week 24 | 78.8 (195.3)
  Change at Week 36: number analyzed (Participants) | 363
  Change at Week 36 | 95.8 (214.4)
  Change at Week 48: number analyzed (Participants) | 344
  Change at Week 48 | 107.4 (213.2)
  Change at Week 60: number analyzed (Participants) | 315
  Change at Week 60 | 131.0 (247.7)
  Change at Week 72: number analyzed (Participants) | 300
  Change at Week 72 | 125.3 (216.1)
  Change at Week 84: number analyzed (Participants) | 266
  Change at Week 84 | 142.8 (223.9)
  Change at Week 96: number analyzed (Participants) | 265
  Change at Week 96 | 143.3 (207.0)
  Change at Week 108: number analyzed (Participants) | 233
  Change at Week 108 | 155.3 (219.8)
  Change at Week 120: number analyzed (Participants) | 219
  Change at Week 120 | 170.9 (233.0)
  Change at Week 132: number analyzed (Participants) | 212
  Change at Week 132 | 180.3 (243.3)
  Change at Week 144: number analyzed (Participants) | 212
  Change at Week 144 | 190.0 (252.9)

4. Secondary Outcome: Percentage of Participants Achieving Absolute CD4 Cell Count Increases From Baseline of ≥ 100 Cells/μL at All Time Points, Modified Intent-to-Treat Analysis
Description: Changes in participants' CD4 cell counts were assessed by measuring the number of CD4 cells at scheduled visits planned as part of routine care.
Time Frame: Baseline (Week 0) to Week 144
Population: Modified 'intent-to-treat' analysis: missing values were replaced by the last observed value of that variable (last observation carried forward method).
Measure: Number; unit: percentage of participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 501
percentage of participants
  Week 4 | 23.8
  Week 12 | 36.5
  Week 24 | 45.7
  Week 36 | 53.1
  Week 48 | 58.1
  Week 60 | 62.7
  Week 72 | 65.1
  Week 84 | 67.7
  Week 96 | 70.5
  Week 108 | 72.3
  Week 120 | 72.5
  Week 132 | 73.1
  Week 144 | 73.7

5. Secondary Outcome: Percentage of Participants Achieving Absolute CD4 Cell Count Increases From Baseline of ≥ 100 Cells/μL at All Time Points, As Treated Analysis
Description: as for outcome 4
Time Frame: Baseline (Week 0) to Week 144
Population: 'As treated' analyses: participants with an assessment, missing data excluded. Number analyzed=participants with an assessment at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 501
percentage of participants
  Week 4: number analyzed (Participants) | 369
  Week 4 | 32.2
  Week 12: number analyzed (Participants) | 400
  Week 12 | 32.5
  Week 24: number analyzed (Participants) | 414
  Week 24 | 37.9
  Week 36: number analyzed (Participants) | 363
  Week 36 | 43.8
  Week 48: number analyzed (Participants) | 344
  Week 48 | 48.0
  Week 60: number analyzed (Participants) | 315
  Week 60 | 50.5
  Week 72: number analyzed (Participants) | 300
  Week 72 | 50.3
  Week 84: number analyzed (Participants) | 266
  Week 84 | 54.5
  Week 96: number analyzed (Participants) | 265
  Week 96 | 55.8
  Week 108: number analyzed (Participants) | 233
  Week 108 | 60.1
  Week 120: number analyzed (Participants) | 219
  Week 120 | 58.0
  Week 132: number analyzed (Participants) | 212
  Week 132 | 58.0
  Week 144: number analyzed (Participants) | 212
  Week 144 | 61.3

6. Secondary Outcome: Time to CD4 Cell Count Increase From Baseline of ≥ 100/ Cells/μL
Time Frame: From Week 0 to Week 144
Population: Participants with an assessment
Measure: Mean (Standard Error); unit: weeks
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 498
weeks | 56.1 (2.8)

7. Secondary Outcome: Number of Participants With Lopinavir (LPV) Resistance at Baseline
Description: Characterization of baseline resistance and development of resistance using the interpretation system HIV-Genotypic Resistance-Algorithm Deutschland (GRADE; available at www.hiv-grade.de.
  Genotypic interpretation was performed using the HIV-GRADE algorithm updated in December 2015). "Susceptible" indicates full susceptibility of a virus to a certain drug without any limitations in terms of resistance. "Partial" resistance is indicated if severe limitations in susceptibility have to be expected and the drug can not count for a fully active drug any more. However, these drugs can still be very useful in situations with generally limited options (salvage). "Resistant" indicates that high level drug resistance has to be expected.
Time Frame: Baseline (Week 0)
Population: Participants with an assessment at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 159
Participants
  Susceptible | 155
  Resistance/Partial Resistance | 4

8. Secondary Outcome: Number of Participants With LPV Resistance During Follow-Up
Description: Characterization of baseline resistance and development of resistance using the interpretation system HIV-GRADE (available at www.hiv-grade.de. Genotypic interpretation was performed using the HIV-GRADE algorithm updated in December 2015). "Susceptible" indicates full susceptibility of a virus to a certain drug without any limitations in terms of resistance. "Partial" resistance is indicated if severe limitations in susceptibility have to be expected and the drug can not count for a fully active drug any more. However, these drugs can still be very useful in situations with generally limited options (salvage). "Resistant" indicates that high level drug resistance has to be expected.
Time Frame: up to Week 144
Population: Participants with an assessment during follow-up; since this was an observational study, resistance testing was performed at the discretion of the treating physician.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 6
Participants
  Susceptible | 5
  Resistance/Partial Resistance | 1

9. Secondary Outcome: Number of Participants With Protease Inhibitor (PI) Resistance at Baseline
Description: as for outcome 7
Time Frame: Baseline (Week 0)
Population: Participants with an assessment at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 159
Participants
  Susceptible | 142
  Resistance/Partial Resistance | 17

10. Secondary Outcome: Number of Participants With PI Resistance During Follow-Up
Description: as for outcome 8
Time Frame: Up to Week 144
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 6
Participants
  Susceptible | 5
  Resistance/Partial Resistance | 1

11. Secondary Outcome: Number of Participants With INI Resistance at Baseline
Description: as for outcome 8
Time Frame: Baseline (Week 0)
Population: Participants with an assessment at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 9
Participants
  Susceptible | 8
  Resistance/Partial Resistance | 1

12. Secondary Outcome: Number of Participants With INI Resistance During Follow-Up
Description: as for outcome 8
Time Frame: up to Week 144
Population: Participants with an assessment at follow-up (neither had available Baseline testing); since this was an observational study, resistance testing was performed at the discretion of the treating physician.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 2
Participants
  Susceptible | 0
  Resistance/Partial Resistance | 2

13. Secondary Outcome: Number of Participants With NNRTI Resistance at Baseline
Description: as for outcome 8
Time Frame: Baseline (Week 0)
Population: Participants with an assessment at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 159
Participants
  Susceptible | 113
  Resistance/Partial Resistance | 46

14. Secondary Outcome: Number of Participants With NNRTI Resistance During Follow-Up
Description: as for outcome 8
Time Frame: up to Week 144
Population: Participants with an assessment at follow-up; since this was an observational study, resistance testing was performed at the discretion of the treating physician.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 6
Participants
  Susceptible | 5
  Resistance/Partial Resistance | 1

15. Secondary Outcome: Number of Participants With Nucleoside Analog Reverse-Transcriptase Inhibitor (NRTI) Resistance at Baseline
Description: as for outcome 8
Time Frame: Baseline (Week 0)
Population: Participants with an assessment at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 159
Participants
  Susceptible | 96
  Resistance/Partial Resistance | 63

16. Secondary Outcome: Number of Participants With NRTI Resistance During Follow-Up
Description: as for outcome 8
Time Frame: up to Week 144
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 6
Participants
  Susceptible | 4
  Resistance/Partial Resistance | 2

17. Secondary Outcome: Number of Participants With HIV-1 Coreceptor Tropism at Baseline
Description: Participants with CCR5 tropic virus, CXC motif chemokine receptor 4 (CRCX4) tropic virus, or dual/mixed tropic virus at Baseline.
Time Frame: Baseline (Week 0)
Population: Participants with an assessment at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 108
Participants
  CCR5 tropic | 74
  CRCX4 tropic | 21
  Dual/mixed tropic | 13

18. Secondary Outcome: Number of Participants With HIV-1 Coreceptor Tropism During Follow-up
Description: Participants with CCR5 tropic virus, CXC motif chemokine receptor 4 (CRCX4) tropic virus, or dual/mixed tropic virus at Follow-up.
Time Frame: up to Week 144
Population: Since this was an observational study, resistance testing was performed at the discretion of the treating physician. No follow-up data on tropism was collected.
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: Change From Baseline in HIV-1 Ribonucleic Acid (RNA) Viral Load
Description: Changes in participants' HIV-1 RNA viral load were assessed by measuring the change from Baseline at scheduled visits planned as part of routine care.
Time Frame: Baseline (Week 0) to Week 144
Population: Participants with an assessment at Baseline. Number analyzed=participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: log copies/mL
Groups:
- HIV-infected Participants: HIV-infected participants on Kaletra and integrase inhibitors or non nucleoside reverse transcriptase inhibitors or CCR5 antagonists
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 500
log copies/mL
  Change at Week 4: number analyzed (Participants) | 389
  Change at Week 4 | -1.37 (1.40)
  Change at Week 12: number analyzed (Participants) | 408
  Change at Week 12 | -1.53 (1.63)
  Change at Week 24: number analyzed (Participants) | 413
  Change at Week 24 | -1.45 (1.70)
  Change at Week 36: number analyzed (Participants) | 367
  Change at Week 36 | -1.49 (1.69)
  Change at Week 48: number analyzed (Participants) | 347
  Change at Week 48 | -1.46 (1.68)
  Change at Week 60: number analyzed (Participants) | 320
  Change at Week 60 | -1.27 (1.62)
  Change at Week 72: number analyzed (Participants) | 304
  Change at Week 72 | -1.32 (1.65)
  Change at Week 84: number analyzed (Participants) | 269
  Change at Week 84 | -1.34 (1.64)
  Change at Week 96: number analyzed (Participants) | 265
  Change at Week 96 | -1.36 (1.59)
  Change at Week 108: number analyzed (Participants) | 233
  Change at Week 108 | -1.32 (1.67)
  Change at Week 120: number analyzed (Participants) | 225
  Change at Week 120 | -1.29 (1.73)
  Change at Week 132: number analyzed (Participants) | 213
  Change at Week 132 | -1.33 (1.65)
  Change at Week 144: number analyzed (Participants) | 216
  Change at Week 144 | -1.38 (1.68)

20. Other Pre Specified Outcome: Time to Virologic Failure
Description: Time to virologic failure was defined by the earliest occurrence of:
  1. HIV-1 RNA > 400 copies/mL confirmed on 2 consecutive occasions after achieving at least 1 HIV-1 RNA < 50 copies/mL,
  2. HIV-1 RNA > 400 copies/mL at the final on-study visit if the participant had previously experienced at least 1 HIV-1 RNA < 50 copies/mL but subsequently did not have HIV-1 RNA > 400 copies/mL on 2 consecutive occasions, or
  3. Day 1 if the participant never achieved HIV-1 RNA < 50 copies/mL during study participation.
  A participant who prematurely discontinued study drug with HIV-1 RNA < 50 copies/mL was censored from analysis at the time of discontinuation provided that he/she did not previously experience either (a), (b) or (c).
Time Frame: Baseline (Week 0) to Week 144
Population: Participants with an assessment
Measure: Mean (Standard Error); unit: weeks
Arm/Group | HIV-infected Participants
Number analyzed (Participants) | 499
weeks | 194.4 (6.2)

ADVERSE EVENTS:
Time Frame: Up to Week 144
Description: Serious adverse events only were collected and coded by MedDRA. Per protocol, the number of participants with events were collected for each event, but from the source documentation to tell how many of the participants are counted in more than one adverse event (i.e., it is not possible to compute the Total Number of Participants Affected). Please see Outcome Measures 1 and 2 for these data.
Arm/Group | HIV-infected Participants
Serious Adverse Events (participants affected / at risk) | 30/501
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-infected Participants (N=501)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 4
NAUSEA (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
FATIGUE (General disorders) | 1
MULTI-ORGAN FAILURE (General disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 1
PYREXIA (General disorders) | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1
AIDS DEMENTIA COMPLEX (Infections and infestations) | 1
ACUTE HEPATITIS C (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 1
CHLAMYDIAL INFECTION (Infections and infestations) | 1
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
INJECTION SITE ABSCESS (Infections and infestations) | 1
LYMPHOGRANULOMA VENEREUM (Infections and infestations) | 1
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
PNEUMONIA FUNGAL (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1
TUBERCULOSIS (Infections and infestations) | 1
YERSINIA INFECTION (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1
ACTINOMYCES TEST POSITIVE (Investigations) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2
INFLAMMATORY MARKER INCREASED (Investigations) | 1
STREPTOCOCCUS TEST POSITIVE (Investigations) | 1
TROPONIN INCREASED (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2
METABOLIC DISORDER (Metabolism and nutrition disorders) | 1
FASCIITIS (Musculoskeletal and connective tissue disorders) | 1
FISTULA (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BUSCHKE-LOWENSTEIN'S TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1
CAROTID ARTERY ANEURYSM (Nervous system disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1
CAROTID ARTERY THROMBOSIS (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DEMENTIA (Nervous system disorders) | 1
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1
SEIZURE (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
VERTEBRAL ARTERY STENOSIS (Nervous system disorders) | 1
WHITE MATTER LESION (Nervous system disorders) | 1
ACUTE PSYCHOSIS (Psychiatric disorders) | 1
DELUSION (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 1
ARTERIAL STENOSIS (Vascular disorders) | 1
ARTERIOSCLEROSIS (Vascular disorders) | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.